CLINICAL TRIAL: NCT06658223
Title: Effects of Immersive Virtual Reality on Quality of Life, Stress, Anxiety, Depression and Cortisol in Fibromyalgia
Brief Title: Effects of Immersive Virtual Reality in Fibromyalgia
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad San Sebastián (Other)
Responsible Party: Principal Investigator, gonzalo arias alvarez, Mrs, Universidad San Sebastián
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3
Record Dates: First submitted 2024-10-23; First posted 2024-10-26 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2024-10

CONDITIONS: Fibromyalgia (FM)
Keywords: FIBROMYALGIA; VIRTUAL REALITY; EXERGAME; EXERCISE
MeSH Terms: conditions — Fibromyalgia; Motor Activity | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Longitudinal quasi-experimental study. The application of the study protocol will be carried out, in its entirety, at the kinesiology center of the Universidad San Sebastián, Concepción campus.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Exercise with virtual reality (Experimental): The virtual reality program consisted of twelve sessions (2 per week for six weeks) of 10 min warm-up plus 15 minutes of exercise with the FitXR game (developed by FITAR LIMITED) on the Oculus Quest 2™ device. The warm-up consisted of moderate-intensity aerobic exercise on a cycle ergometer. The BORG CR-10 perceived exertion scale was used to determine this intensity. Subsequently, they continued with the FitXR game, starting with a 5-minute phase of muscular activation and global movements of their limbs. They performed eye-hand coordination exercises, hitting balls that came to the person at different speeds, and ended with muscle stretching and slow breathing. These exercises presented different difficulty levels and were adjusted to the person's condition. In the same way, as the game developed, it was possible to increase the level and thus increase its complexity.
  Interventions: Other: Exercise with virtual reality

INTERVENTIONS:
Other: Exercise with virtual reality — The virtual reality program consisted of twelve sessions (2 per week for six weeks) of 10 min warm-up plus 15 minutes of exercise with the FitXR game (developed by FITAR LIMITED) on the Oculus Quest 2™ device. The warm-up consisted of moderate-intensity aerobic exercise on a cycle ergometer. The BORG CR-10 perceived exertion scale was used to determine this intensity. Subsequently, they continued with the FitXR game, starting with a 5-minute phase of muscular activation and global movements of their limbs. They performed eye-hand coordination exercises, hitting balls that came to the person at different speeds, and ended with muscle stretching and slow breathing. These exercises presented different difficulty levels and were adjusted to the person's condition. In the same way, as the game developed, it was possible to increase the level and thus increase its complexity.

SUMMARY:
Fibromyalgia is considered a disease of unknown etiology, which It affects between 2 to 5% of the population in developed countries, mostly women, diagnosed mainly between 40 and 50 years of age, and whose main characteristic is generalized presence of musculoskeletal pain. Although the most described symptoms are multiple sensitive areas in trigger points, fatigue and cognitive dysfunction, this syndrome is associated commonly to anxiety disorders, depression and catastrophizing. In Chile, consultations specific cases of rheumatology due to Fibromyalgia reach 26.7%, with a similar reality in the commune of Concepción, as a result of which the need arises to implement a strategy different and innovative, in which an environment can be generated in which the user practices motor and cognitive strategies in different contexts, whether work or home, to through virtual reality, which has proven to be a promising tool in this group of the population, since by entering a controlled virtual environment, different techniques, taking them out of the conventional treatment box. In this way, it may include relaxation exercises, cognitive behavioral therapy, and physical activities adapted. This interaction may improve cognitive function, reduce anxiety symptoms, reduce painful perception associated with your health condition and improve your quality of life. Although there is knowledge and favorable experiences in its use, there is little information about the effects and the scope that it can have in patients with fibromyalgia. For this reason, it is proposed to carry out an investigation applying a Kinesiological treatment complemented with virtual reality. in patients with this disease. Therefore, the research question arises: What is the effectiveness of a kinesiological treatment, complemented with immersive virtual reality, on quality of life, cognitive and psychoemotional function in patients with fibromyalgia?

DETAILED DESCRIPTION:
According to the World Health Organization (WHO), fibromyalgia is considered a disease of unknown etiology, which affects between 2 and 5% of the population of developed countries, mostly women, diagnosed mainly between the ages of 40 and 50. In Chile, the prevalence is in a range between 1 and 2%. This disease is characterized by persistent generalized musculoskeletal pain, emotional symptoms such as anxiety, depression and cognitive disorders that mainly affect concentration and memory and compromise their quality of life.

It is for this reason that the need arises to implement a different, innovative strategy, in which an environment can be generated in which the patient can put motor and cognitive strategies into practice in different contexts, whether work or home, through virtual reality.

Virtual reality has proven to be a promising tool in the treatment of fibromyalgia. When patients enter a controlled virtual environment, they can work on different techniques that avoid conventional treatment pigeonholing. Current evidence describes the effectiveness of virtual reality in chronic pain syndromes, rheumatoid arthritis and especially in central neurological injuries, incorporating relaxation exercises and adapted physical activities. This interaction can improve cognitive function and reduce symptoms of anxiety and depression associated with their health condition. Although there is favorable knowledge and experiences in its use, there is little information about the effects and scope that it can have in patients with fibromyalgia, which is why it is proposed to carry out research applying a Kinesiological treatment complemented with virtual reality in patients with this disease. Therefore, the research question arises: What is the effectiveness of a kinesiological treatment, complemented with immersive virtual reality, on quality of life, cognitive and psychoemotional function in patients with fibromyalgia?

ELIGIBILITY:
Inclusion Criteria:

* Males and females
* over 18 years of age
* with a diagnosis of fibromyalgia issued by a medical professional under the ACR criteria (2016)

Exclusion Criteria:

* Subjects were excluded from the study when they presented pregnancy or lactation
* oncologic pain
* uncontrolled metabolic disorder
* vertigo or similar condition or any cognitive impairment that hinders the understanding of the informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-09-02 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-02-28 (Estimated)

PRIMARY OUTCOMES:
Impact of Fibromyalgia on Quality of Life | SIX WEEKS
  The Impact of Fibromyalgia on Quality of Life was assessed using the FIQ-R instrument. This self-administered test measures difficulty in activities of daily living in the last week, the overall influence of the disease in the last week, and the severity of symptoms in the past week. Total scores range from 0 to 100, with higher scores indicating more severe symptoms and disability.

SECONDARY OUTCOMES:
Cortisol | SIX WEEKS
  Cortisol levels will be measured using the Cortisol ELISA saliva kit from the manufacturer IBL International Gmbh ®. Prior to the experiment, subjects will be asked not to consume solid or liquid food 60 minutes before the test, as recommended by the manufacturer. The sample collection procedure will be carried out according to the manufacturer's guidelines. They will then be stored at -20°C until the respective analysis is carried out. The sample will be kept away from heat and direct sunlight. The entire procedure will be carried out in the laboratories of the Medical Technology Department of the Universidad San Sebastián, Concepción campus.
Stress, anxiety and depression | SIX WEEKS
  Stress, anxiety, and depression were assessed using the Depression Anxiety Stress Scale-21 (DASS-21). This self-administered dimensional test consists of twenty-one questions to evaluate three categories, specifically stress, anxiety, and depression. It presents four response options for each category, evaluated on a scale from 0 to 3. The score obtained for each category is multiplied by 2, and the result is classified as normal, mild, moderate, severe, and extremely severe.
Cognitive function | SIX WEEKS
  Cognitive function in both groups will be assessed by applying the MoCA questionnaire, a brief cognitive assessment test that measures the performance of abilities such as memory, orientation, language, concentration, executive function and visuospatial skills.

CONTACTS AND LOCATIONS:
Overall Officials: GONZALO J ARIAS-ALVAREZ, Principal Investigator — Universidad San Sebastián
Locations (1):
- Universidad San Sebastián, Concepción, Bio-bio, Chile

IPD SHARING:
Plan to Share IPD: Undecided
WE ARE NOT SURE ABOUT IT, BUT WE DO NOT REFUSE TO GRANT IT LATER ON.